CLINICAL TRIAL: NCT06693986
Title: A Phase I Study of a Tropism Modified Conditionally Replicative Adenovirus Vector (RGDCRAdCOX2F) for Endoscopic, Direct-Tumor Delivery in Pancreatic Adenocarcinoma
Brief Title: Adenovirus (RGDCRAdCOX2F)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022LS030
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma of Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Level: -1 RGDCRAdcox2F (RGD) (Experimental): Patients given 3x10^10 vp/d of RGD.
  Safety arm. Enrollment begins at DL 1 in cohorts of 2 patients. A minimum of 28 days (DLT period) must separate the last patient treated in the current cohort and the 1st patient in the next cohort of 2 patients. A minimum of 21 days must separate the 1st and 2nd patient within a cohort.
  Interventions: Biological: Replicative Adenovirus Vector (RGDCRAdCOX2F)
- Level: 1 RGDCRAdcox2F (RGD) (Experimental): Patients given 3x10^11 vp/d of RGD
  Enrollment begins at DL 1 in cohorts of 2 patients. A minimum of 28 days (DLT period) must separate the last patient treated in the current cohort and the 1st patient in the next cohort of 2 patients. A minimum of 21 days must separate the 1st and 2nd patient within a cohort.
  Interventions: Biological: Replicative Adenovirus Vector (RGDCRAdCOX2F)
- Level: 2 RGDCRAdcox2F (RGD) (Experimental): Patients given 9x10^11 vp/d of RGD.
  Enrollment begins at DL 1 in cohorts of 2 patients. A minimum of 28 days (DLT period) must separate the last patient treated in the current cohort and the 1st patient in the next cohort of 2 patients. A minimum of 21 days must separate the 1st and 2nd patient within a cohort.
  Interventions: Biological: Replicative Adenovirus Vector (RGDCRAdCOX2F)
- Level: 3 RGDCRAdcox2F (RGD) (Experimental): Patients given 3x10^12 vp/d of RGD.
  Enrollment begins at DL 1 in cohorts of 2 patients. A minimum of 28 days (DLT period) must separate the last patient treated in the current cohort and the 1st patient in the next cohort of 2 patients. A minimum of 21 days must separate the 1st and 2nd patient within a cohort.
  Interventions: Biological: Replicative Adenovirus Vector (RGDCRAdCOX2F)

INTERVENTIONS:
Biological: Replicative Adenovirus Vector (RGDCRAdCOX2F) — RGDCRAdcox2F (RGD) is a "local" product and is provided through this study.

SUMMARY:
This is a single center, Phase I dose finding study of a single direct tumor injection of an RGD modified conditionally replicative adenovirus (RGDCRAdcox2F) in persons with adenocarcinoma of the pancreas. The study is designed to determine the MTD of RGDCRAdCOX2F that corresponds to the maximum desired toxicity of ≤ 20%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented pancreatic adenocarcinoma that is confined to the pancreas and regional lymph nodes after staging by CT or MRI and endoscopic ultrasound.
* One prior line of therapy is permitted (i.e. neo-adjuvant therapy); however, at least 4 weeks must have elapsed between the last dose of drug and the injection of RGDCRAdCOX2F.
* Must be able to tolerate esophagogastroduodenoscopy (EGD) and the tumor must be accessible by endoscopic ultra sound. Participants will be excluded if obtaining biopsies are deemed unsafe or not feasible.
* Age 18 years of age or older at the time of consent
* Normal cardiac and pulmonary function based on history and physical exam
* Participants with partners of childbearing potential must be willing to use at least two forms of effective birth control (one form must be a barrier method) for at least 1 month after Day 1.

Exclusion Criteria:

* Pregnant or breastfeeding. Persons of child-bearing potential must have a negative pregnancy test (serum or urine) with 14 days of study enrollment.
* Other pancreatic malignancies (e.g., neuroendocrine tumors and mucinous cystic) and adenocarcinomas of the ampulla, bile ducts, and duodenum.
* Tumors in mucosal regions or close to an airway, major blood vessel, or spinal cord that in the opinion of the enrolling investigator could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis.
* Known history of human immunodeficiency virus (HIV) infection
* Known history of or active acute or chronic active hepatitis B or C infection
* Serious concurrent infection or medical illness, which in the enrolling investigator's opinion would jeopardize the ability of the participant to receive the treatment outlined in this protocol with reasonable safety.
* Requires immunosuppression ≥10mg/day of prednisone for more than

  1 week.
* History of or active known or suspected autoimmune disease, or a syndrome that requires systemic or immunosuppressive agents.
* Disease beyond the regional lymph nodes
* Active diffuse pancreatitis
* Active inflammatory conditions
* Prior gastrojejunostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose Limiting Toxicity (DLT) Events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States